CLINICAL TRIAL: NCT05292911
Title: A 12-Week Extension Study of ALT-801 in Diabetic and Non-Diabetic Overweight and Obese Subjects With Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Extension of ALT-801 in Diabetic and Non-Diabetic Overweight and Obese Subjects With (NAFLD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-801-106
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Obese; Overweight
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Overweight | interventions — ALT-801

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALT-801 Dose Level 1 (Experimental): Administered once a week for 12 weeks
  Interventions: Drug: ALT-801
- ALT-801 Dose Level 2 (Experimental): Administered once a week for 12 weeks
  Interventions: Drug: ALT-801
- ALT-801 Dose Level 3 (Experimental): Administered once a week for 12 weeks
  Interventions: Drug: ALT-801
- Placebo (Placebo Comparator): Administered once a week for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ALT-801 — Injected subcutaneously (SC)
  Other Names: Pemvidutide
  Arms: ALT-801 Dose Level 1; ALT-801 Dose Level 2; ALT-801 Dose Level 3
Other: Placebo — Injected subcutaneously (SC)
  Arms: Placebo

SUMMARY:
This extension study will assess the safety and effects of 24 weeks of treatment with ALT-801 in diabetic and non-diabetic subjects with overweight and obesity and non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
This extension study will enroll subjects who have completed 12 weeks of treatment in Study ALT-801-105. It is designed to allow for an additional 12 weeks of treatment in order to assess the safety and effects of 24 weeks of treatment with ALT-801 in diabetic and non-diabetic subjects with overweight and obesity and non-alcoholic fatty liver disease (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this extension study, signed prior to the performance of any study procedures
* Receipt of 12 weeks of investigational product with completion of the procedures in Study ALT-801-105
* Women who are not pregnant or breastfeeding

Exclusion Criteria:

* Meets any of the exclusion criteria in Study ALT-801-105 at the time of study entry
* Development of any of the following conditions at any time during Study ALT-801-105:

  1. Type 1 DM and/or insulin-dependent type 2 diabetes mellitus (T2DM), or uncontrolled T2DM requiring rescue therapy in study ALT-801-105
  2. History of pancreatitis or hypersensitivity reaction to GLP-1 analogues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) | Up to Day 110
  Number of participants with one or more TEAEs

SECONDARY OUTCOMES:
Change from baseline in liver fat fraction by MRI-PDFF | Baseline to Day 85
  Change in MRI-PDFF
Change from baseline in body weight | Baseline to Day 85
  Change in body weight
Change from baseline in lipid metabolism (total cholesterol, HDL cholesterol, LDL cholesterol, lipoprotein fractions) | Baseline to Day 85
  Change in lipid metabolism (TC, HDL, LDL)
Change from baseline in hemoglobin A1c | Baseline to Day 85
  Change in hemoglobin A1c
Change from baseline in fibrosis markers (Pro-C3) | Baseline to Day 85
  Change in fibrosis markers (Pro-C3)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Browne, MD, Study Director — Altimmune, Inc.
Locations (13):
- United States (13):
  - Catalina Research Institute, Montclair, California
  - Clinical Trials Research, Sacramento, California
  - Panax Clinical Research, Miami Lakes, Florida
  - Covenant Research and Clinics, Sarasota, Florida
  - Headlands Research Sarasota, Sarasota, Florida
  - Wake Research CRCN, Las Vegas, Nevada
  - Accelemed Research Institute, Austin, Texas
  - Pinnacle Research, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Pinnacle Research, San Antonio, Texas
  - Cognitive Clinical Trials, Salt Lake City, Utah

REFERENCES:
- [Derived] Browne SK, Suschak JJ, Tomah S, Gutierrez JA, Yang J, Georges B, Roberts MS, Harris MS. Safety and efficacy of 24 weeks of pemvidutide in metabolic dysfunction-associated steatotic liver disease: A randomized, controlled clinical trial. JHEP Rep. 2025 Jun 18;7(11):101483. doi: 10.1016/j.jhepr.2025.101483. eCollection 2025 Nov. PMID 41113119